CLINICAL TRIAL: NCT06639594
Title: Feasibility of Accelerated, Personalized rTMS as an Adjuvant for Impulse Control Disorders: a Pilot Study
Acronym: RAPID
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0261; NCI-2024-08561 (Other: NCI CTRP Clinical Registry)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Impulse Control Disorder
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intermittent theta burst stimulation (Experimental): Participants undergo rTMS once a week for 2 weeks. In week 1 participants receive continuous theta burst stimulation (cTBS) for 3 sessions; in week 2 participants receive intermittent theta burst stimulation (iTBS) for 3 sessions. Additionally, participants complete cued food delivery task assessment and undergo saliva sample collection on study.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Continuous theta burst stimulation (Experimental): Participants undergo rTMS once a week for 2 weeks. In week 1 participants receive continuous theta burst stimulation (cTBS) for 3 sessions; in week 2 participants receive intermittent theta burst stimulation (iTBS) for 3 sessions. Additionally, participants complete cued food delivery task assessment and undergo saliva sample collection on study.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — RTMS is a non-invasive procedure in which a coil is placed over the scalp, and powerful, focused magnetic pulses are applied to parts of the brain through the coil.

SUMMARY:
To learn if accelerated rTMS (repetitive transcranial magnetic stimulation) can be used as a possible therapy for excessive eating.

DETAILED DESCRIPTION:
Primary Objectives:

To evaluate the feasibility of using accelerated rTMS as a potential treatment adjuvant, we will assess the following feasibility primary outcomes:

-Recruitment: We will define recruitment as the probability of an eligible participant consenting to participate in the study.

We will deem recruitment for this trial feasible if at least 70% of eligible participant consent to participate in the trial. (i.e., considering a pool of 30 eligible participant, we consent at least 21 participants).

* Tolerability: For each protocol, we will follow an up-titration procedure (from 80% up to 110% of the motor threshold) and define the optimally tolerable dose (OTD) as the dose that at least 70% of participants can tolerate. Tolerability will be computed separately for each rTMS protocol.
* Safety: To consider the treatment safe, there must be no serious adverse events attributable to rTMS.

Secondary Objectives

We will measure:

1. To measure the time required to the staff to conduct each ERP assessment.
2. To measure the time between the end of the last rTMS session and the start of the second ERP assessment.

   We will analyze each measure to obtain an accurate estimate of the duration of each step in the procedures. Our ultimate goal is to develop image-guided, personalized rTMS interventions. Carefully assessing the time required for each step in the protocol will allow us to identify opportunities to further optimize our procedures and reduce the duration of future visits.
3. We will conduct exploratory analyses on the amplitude of the late positive potential (LPP) component of the ERPs. Our exploratory analyses will allow us to estimate the LPP responses collected from the "cued food delivery task" before and after the rTMS intervention and assess the level of noise in the data by computing the standardized measurement error (SME).

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 to 60
2. BMI>30 (confirmed at in person visit)
3. Able to follow verbal and written instructions in English and complete all aspects of the study.
4. Have an address and telephone number where they may be reached.
5. Subjects must report current stable residence. Stable residence is a domicile in which an individual can operate as if it were their own homestead and does not include shelters, halfway houses, treatment centers, or group homes.
6. Meet safety criteria for EEG and rTMS.
7. Willing and able to independently remove any metal from the neck and above for rTMS procedures (e.g., jewelry, retainer)
8. Provides written informed consent and agree to all assessments and study procedures.
9. Agrees to complete telehealth (live audio-video conference and phone) and in-person visits and to be contacted via text.

Exclusion Criteria

1. rTMS exposure for treatment or research purposes in the last 6 months.
2. History of seizure, epilepsy, syncope, fainting episode, or head trauma resulting in loss of consciousness.
3. Presence or history of neurological disorders (migraine, stroke, Alzheimer's Disease and other Dementias, Parkinson's Disease, Multiple Sclerosis, Traumatic Brain Injury (TBI), increased intracranial pressure).
4. History of brain surgery, implanted electronic device, metal in the head.
5. Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps or sensors, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes)
6. History of or currently under medical care for myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke, or transient ischemic attack.
7. Reported history of vision problems that are not treated.
8. Has a hairstyle not compatible with the EEG net that is required to be worn on the scalp during the experimental procedure.
9. Reports current diagnosis or history of type I diabetes.
10. Currently using insulin.
11. Have undergone bariatric surgery.
12. Currently being enrolled in a weight loss program
13. Takes any prescription or over the counter medications or supplements to control weight and/or appetite.
14. Self-report a history of or current diagnosis of a mental health condition.
15. Reports insomnia (<4 hours sleep per night, in 3 or more nights per week in the last 3 months)
16. Reports (<4 hours of sleep) the day of the visit.
17. Reports using marijuana on a daily basis.
18. Reports having used any other illicit drugs (other than marijuana) or prescription medications for non-medical reasons in the last 12 months.
19. Currently receiving treatment for substance use disorder (e.g., alcohol, opioids, cocaine, marijuana, or stimulants).
20. Females who report averaging more than 7 alcoholic drinks, or males who report averaging more than 14 alcoholic drinks in a single week in the last 30 days.
21. Current use of certain medications (last 3 months):

    * Investigational drugs.
    * Drugs of anti or pro-convulsive action. Medications with psychotropic effects (e.g., antidepressants, antipsychotics).
    * Medications known to increase risk of seizure taken within 1 week of enrollment.
    * Smoking cessation medication (e.g., Zyban, Wellbutrin, Wellbutrin SR, Chantix).
22. Being pregnant or lactating
23. Reported allergies to chocolate or any ingredient in the M&M candies.
24. Noise-induced hearing loss or tinnitus.
25. Currently participating in any other research study.
26. Any otherwise not specified medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician
27. Subjects considered by the investigator as unsuitable for the study for reasons not otherwise stated.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2027-11-03 (Estimated); Study Completion 2027-11-03 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs). | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Versace, PHD,PHD, Principal Investigator — The Unversity of Texas MD Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org